CLINICAL TRIAL: NCT02966041
Title: A Double-blinded, Randomized Control Trial of Prophylactic Ondansetron in a Post-operative Cardiac Surgery Population for Post-operative Nausea and Vomiting
Brief Title: Prophylactic Ondansetron in Post-op Cardiac Surgery Patients to Prevent Post-operative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Matthew Coley, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H15-00675
Record Dates: First submitted 2016-10-25; First posted 2016-11-17 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; PONV; CSICU; post-cardiac surgery; cardiac intensive care unit
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron (Experimental): Ondansetron 4mg IV at time of discontinuation of Propofol Infusion
  Interventions: Drug: Ondansetron
- Saline (Placebo Comparator): 2 mL IV Normal Saline at time of discontinuation of Propofol Infusion
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ondansetron — Ondansetron/Zofran is an antiemetic drug used to prevent and treat nausea and vomiting.
  Other Names: Zofran
  Arms: Ondansetron
Drug: Saline — Normal saline is salt water and is acting as a placebo in this study. A placebo is an inactive substance that looks identical to the test drug, but it contains no therapeutic ingredient.
  Other Names: Placebo Comparator: Saline
  Arms: Saline

SUMMARY:
To evaluate the effectiveness of a prophylactic dose of ondansetron in decreasing the incidence of post-operative nausea and vomiting in cardiac surgery patients after cessation of post-operative sedation. In patients who have undergone open heart surgery, a single prophylactic dose of ondansetron 4 mg IV given at the time of discontinuing propofol sedation will result in a 50% reduction of the rate of post-operative nausea and vomiting in the first 24 post-operative hours compared to placebo.

DETAILED DESCRIPTION:
Post-operative nausea and vomiting (PONV) is a significant source of morbidity for patients undergoing general anesthesia, and in particular, patients undergoing cardiac anesthesia. Despite its common occurrence, literature on PONV prophylaxis in the cardiac surgical population is limited relative to other surgical populations.

A rational approach to preventing PONV would be to administer prophylaxis prior to extubation once post-operative sedation has ceased. This timing of administration would be more standardized across patients, as duration of surgery and time of extubation after surgery can vary considerably, rendering plasma levels of PONV prophylaxis agents highly variable across patients.

At St. Paul's Hospital, PONV prophylaxis has not been a routine part of cardiac anesthesia care. Furthermore, there are no standardized guidelines, and practice varies between care providers. Following surgery, patients recover from anesthesia and are extubated in the cardiac surgery ICU (CSICU). They are usually sedated on a propofol infusion for one to four hours after surgery until they are ready for extubation. When PONV occurs, the first line drug for treatment is ondansetron 4 mg. The investigators therefore propose the use of a single, prophylactic dose of ondansetron (4 mg IV), given at the time of propofol cessation. A randomized, double blinded placebo controlled model will be utilized

ELIGIBILITY:
Inclusion Criteria:

* Elective (outpatient) and urgent (inpatient) cardiac surgery procedures requiring cardiopulmonary bypass, including:

  * Coronary artery bypass grafting (CABG)
  * Valve surgery (ie. repair and/or replacement)
  * CABG and valve surgery

Exclusion Criteria:

* Undergoing 'off-pump' CABG (not involving the cardiopulmonary bypass machine)
* With a contraindication to the study drug - including but not limited to congenital Long QT Syndrome, allergy to ondansetron, or a history of migraines
* Unable to understand the consent process, either due to language limitations or cognitive limitations if a translator or substitute decision maker is not available
* Receiving heart transplants, ventricular assist devices or on extra-corporeal membrane oxygenation (ECMO)
* Intubated for more than 12 hours post-operatively
* With a known history of PONV
* Sedated with dexmedatomine instead of propofol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of Post-operative Nausea and Vomiting (PONV) | First 24 hours post-extubation
  Measured by asking the patient hourly to assess their post operative nausea and vomiting using a 10-point verbal Likert rating scale.

SECONDARY OUTCOMES:
Incidence of Rescue PONV medication administration | First 24 hours post-extubation
  How many participants received rescue post-operative nausea and vomiting medication post-extubation after surgery.
Time to first dose of rescue PONV medication | First 24 hours post-extubation
  Time of administration of first dose of rescue post-operative nausea and vomiting medication
Dose of any Rescue PONV medication | First 24 hours post-extubation
  Dose of administered rescue post-operative nausea and vomiting medication after extubation.
Time to first report of nausea or first vomit post-operatively | First 24 hours post-extubation
  Time to first report of any nausea or vomiting after extubation post-operatively.
Incidence of Post-operative nausea without vomiting | First 24 hours post-extubation
  Nurses both asked patients' for a nausea severity rating and recorded any vomiting hourly.
Severity Post-operative nausea without vomiting | First 24 hours post-extubation
  Severity of post-operative nausea without vomiting based on a 10-point likert scale, recorded hourly.
Incidence of ventricular arrhythmias | first 24 hours post-extubation
  Any sustained Ventricular Arrhythmias (i.e. lasting greater than 30 seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Coley, MD, Principal Investigator — University of British Columbia; Erica Wang, PharmD, Study Chair — University of British Columbia; Cynthia Yarnold, MD, Study Chair — University of British Columbia; Stephan Schwarz, MD, Study Chair — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang EHZ, Sunderland S, Edwards NY, Chima NS, Yarnold CH, Schwarz SKW, Coley MA. A Single Prophylactic Dose of Ondansetron Given at Cessation of Postoperative Propofol Sedation Decreases Postoperative Nausea and Vomiting in Cardiac Surgery Patients: A Randomized Controlled Trial. Anesth Analg. 2020 Oct;131(4):1164-1172. doi: 10.1213/ANE.0000000000004730. PMID 32925337